CLINICAL TRIAL: NCT01641016
Title: BREATHER (PENTA 16) Short-Cycle Therapy (SCT) (5 Days on/2 Days Off) in Young People With Chronic HIV-infection
Acronym: BREATHER
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: PENTA Foundation (Network)
Collaborators: Medical Research Council (Other Government); ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BREATHER (PENTA 16); 2009-012947-40 (EudraCT Number)
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2015-03-02 (Estimated); Status verified 2013-07

CONDITIONS: HIV
Keywords: short cycle therapy; young people; HIV
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Therapy (Active Comparator): Continue with current antiretroviral therapy regime as per standard care
  Interventions: Drug: efavirenz
- Short Cycle Therapy (Experimental): Take current antiretroviral therapy 5 days a week (2 days off) as instructed by clinician
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: efavirenz — May be taken as 600mg tablet, 200mg tablet or as part of a combination pill
  Other Names: Trade name: Sustiva

SUMMARY:
The overall aim of the BREATHER trial is to evaluate the role of Short-Cycle Therapy (SCT) in the management of HIV-infected young people who have responded well to antiretroviral therapy (ART) and to determine whether young people with chronic HIV infection undergoing Short-Cycle Therapy of five days on ART and two days off maintain the same level of viral load suppression as those on continuous therapy, over 48 weeks.

To assess the advantages and disadvantages of the strategy, the incidence of toxicities, immunological control, resistance mutations, acceptability, quality of life and adherence to the randomised strategy will also be compared.

Importantly, because of insufficient data on short-term viral load rebound after stopping ART in this population, the trial will incorporate an initial pilot phase in selected centres, to assess the safety of the SCT strategy by evaluating detailed HIV-1 RNA profiles of participants on the SCT strategy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected young people aged 8 to 24 years inclusive (Young people recruited between the ages of 16-21 must either be in regular physical contact with their clinician or be able to transfer to an adult physician at the same site for follow-up or to an affiliated adult site).
* Parents/carers and/or young people, where applicable, willing to provide informed consent.
* On a stable first-line ART treatment containing at least 2 NRTIs/NtRTIs and EFV for at least 12 months and willing to continue the regimen throughout the study period. Young people on regimens containing nevirapine (NVP) or a boosted protease inhibitor with undetectable viral load for over one year who wish to enrol should switch to EFV. Once they are stable on the EFV containing regimen for more than 12 weeks they may be enrolled (must have 2 subsequent HIV-1 RNA measurements <50 c/ml over a minimum period of 12 weeks). Previous dual therapy and/or substitution of NRTIs is allowed providing any changes were not for disease progression, immunological or virological failure (where virological failure is defined as two successive HIV-1 RNA results>1000 c/ml) subsequent to virological control having been achieved on ART.
* Viral suppression (HIV-1 RNA <50 c/ml) for at least the prior 12 months (at least the last 3 measurements, including screening): young people who have experienced a single viral load >50 but <1000 copies/ml (preceded and followed by VL<50 c/ml) in the last 12 months can be enrolled.
* CD4 cell count ≥350 106/L at screening visit.
* Centre must routinely use an assay which detects HIV RNA-1 viral load ≥50 c/ml.

Exclusion Criteria:

* Pregnancy or risk of pregnancy in females of child bearing potential.
* Acute illness (young people may be enrolled after illness).
* Receiving concomitant therapy for an acute illness (young people may be enrolled after finishing therapy).
* A creatinine, AST or ALT of grade 3 or above at screening.
* On a regimen including nevirapine or a boosted PI (young people may switch to an EFV based regimen).
* Previous ART monotherapy (except for the prevention of mother-to-child transmission)

Ages: 8 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
HIV-1 RNA ≥50 copies/ml (confirmed on a separate sample within 1 week) at any of week 4, 12, 24, 36 or 48. | 48 weeks
  This outcome measure only considers HIV-1 RNA measurements at these time points due to the difference in viral load monitoring in the pilot phase and the main trial. However if a young person enrolled in the pilot phase has HIV-1 RNA ≥50 copies/ml at weeks 1, 2 or 3 (reproducible on the same sample) or at week 8 (confirmed on the same sample within 1 week), they will be considered as reaching the primary outcome at week 4 and 12 respectively

SECONDARY OUTCOMES:
HIV-1 RNA <50 c/ml at 24 and 48 weeks | 24 and 48 weeks
Number of HIV mutations present at week 4, 12, 24, 36 or 48 conferring resistance to drugs taken at randomisation or during the tria | Weeks 4, 12, 24, 36, 48
Change in CD4 (absolute and percentage) from randomisation to 24 and 48 weeks | 24 and 48 weeks
Change in ART (defined as any change from the ART regimen at randomisation) | 48 weeks
Grade 3 or 4 clinical and laboratory adverse events | 48 weeks
ART treatment modifying adverse events (all grades) | 48 weeks
New CDC stage B or C diagnosis or death | 48 weeks
Changes in fasting glucose, cholesterol, triglycerides, LDL, HDL and VLDL levels through 48 weeks | 48 weeks
Adherence, acceptability, and quality of life over 48 weeks as assessed by patient completed questionnaires | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karina M Butler, MRCPI, Principal Investigator — Medical Research Council
Locations (18):
- St Jude Children's Research Hospital, Memphis, Tennessee, United States
- INSERM, Villejuif, France
- Universitätsklinikum Frankfurt, Frankfurt, Frankfurt Am Main, Germany
- Our Lady's Children's Hospital, Dublin, Ireland
- Thailand (2):
  - Program for HIV Prevention and Treatment (PHPT)/IRD 174, Changklan, Muang, Chiang Mai
  - HIV-NAT Thai Red Cross AIDS Research Centre, Bangkok
- Joint Clinical Research Centre, Kampala, Uganda
- Kiev City AIDS Center, Kiev, Vidpochynku 11, Ukraine
- United Kingdom (10):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospital Bristol, Bristol
  - Leeds General Infirmary, Leeds
  - Leicester Royal Infirmary, Leicester
  - Evelina Children's Hospital, London
  - Great Ormond Street Hospital, London
  - Mortimer Market Centre, London
  - St George's Hospital, London
  - Nottingham University Hospital, Nottingham
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Turkova A, Moore CL, Butler K, Compagnucci A, Saidi Y, Musiime V, Nanduudu A, Kaudha E, Cressey TR, Chalermpantmetagul S, Scott K, Harper L, Montero S, Riault Y, Bunupuradah T, Volokha A, Flynn PM, Bologna R, Ramos Amador JT, Welch SB, Nastouli E, Klein N, Giaquinto C, Ford D, Babiker A, Gibb DM; BREATHER (PENTA 16) trial Group. Weekends-off efavirenz-based antiretroviral therapy in HIV-infected children, adolescents and young adults (BREATHER): Extended follow-up results of a randomised, open-label, non-inferiority trial. PLoS One. 2018 Apr 23;13(4):e0196239. doi: 10.1371/journal.pone.0196239. eCollection 2018. PMID 29684092
- [Derived] Bernays S, Paparini S, Seeley J, Namukwaya Kihika S, Gibb D, Rhodes T. Qualitative study of the BREATHER trial (Short Cycle antiretroviral therapy): is it acceptable to young people living with HIV? BMJ Open. 2017 Feb 17;7(2):e012934. doi: 10.1136/bmjopen-2016-012934. PMID 28213595
- See also: Related Info — http://www.pentatrials.org/